CLINICAL TRIAL: NCT03283852
Title: Identifying New Genetic Causes to the Disorders of Growth, Puberty and Sex Development
Brief Title: Identifying New Genetic Causes to Development Disorders
Acronym: FORDEV
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: RBR_2016_16
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Disorders of Sex Development; Growth Disorders; Puberty Disorders
MeSH Terms: conditions — Disorders of Sex Development; Growth Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — •Samples With DNA: serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: blood sample — search for genetic mutations

SUMMARY:
Disorders of growth, puberty and sex development can have genetic causes. The exome analysis could detect new mutations responsible for these disorders and the frequency of these mutations in these disorders, their association with other malformations.

ELIGIBILITY:
Inclusion Criteria:

* congenital growth hormone deficiency
* puberty disorder
* gonadal dysgenesis or anorchia
* primary ovarian failure
* disorder of sex development
* subjects related to a patient with one of the above criteria

Exclusion Criteria:

* environmental or auto-immune cause

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with disorders of growth, puberty and sex development and related subjects.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2017-02-21 (Actual); Primary Completion 2027-02-21 (Estimated); Study Completion 2027-02-21 (Estimated)

PRIMARY OUTCOMES:
mutation research | baseline
  frequency of genetic mutation

CONTACTS AND LOCATIONS:
Overall Officials: Raja Brauner, PU-PH, Principal Investigator — Hôpital Fondation A. de Rothschild
Locations (1):
- Hôpital Fondation A de Rothschild, Paris, France